CLINICAL TRIAL: NCT06370338
Title: Delphi Study for Evaluation of Cardiothoracic Critical Care as a Subspecialty and Its Core Competencies
Brief Title: Cardiothoracic Critical Care as Subspecialty and Its Core Competencies
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Rafal Kopanczyk, Assistant Professor - Clinical, Ohio State University
Other Study IDs: 2024B0101
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Consensus Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Delphi Panel: Experts in the field of cardiothoracic critical care with administrative, educational, and research roles.
  Interventions: Other: Delphi Questionnaire

INTERVENTIONS:
Other: Delphi Questionnaire — Experts will be approached to participate in the research via email. If the experts agree to participate they will check 'yes' in the email with the informed consent and will be directed to the Qualtrics survey. If the expert decides to decline consent they will check 'no' in the email and will not be enrolled. Subjects who agree to participate will undergo 2 phases of questions with three rounds of the same questions in each phase. This Delphi survey research involves Phase 1 and Phase 2 of questioning, each phase involves up to 3 rounds of questions to determine agreement or disagreement. Each round will take approximately 20 minutes to complete, and your responses will remain completely confidential. For both phases, the questions will either be 7-point Likert or multiple choices. For both phases, the group of questions will be sent up to three times until we obtain agreement (up to 80% of agreement consensus). Questions that have obtained agreement will be removed in each round.

SUMMARY:
The aim of this study is to develop a consensus on the curriculum for training cardiothoracic critical care by first evaluating the need for the field, based on a Delphi consensus among a panel of experts in this field.

DETAILED DESCRIPTION:
This study will use the Delphi process to conduct this study. This survey research involves Phase 1 and Phase 2 of questioning, each phase involves up to 3 rounds of questions to determine agreement or disagreement. Each round will take approximately 20 minutes to complete, and responses will remain completely confidential. For both phases, the questions will either be 7-point Likert or multiple choices. For both phases, the group of questions will be sent up to three times until agreement (up to 80% of agreement consensus). Questions that have obtained agreement will be removed in each round. The questions will help the experts and the research team understand where there is current agreement on, or topic that may need to be discussed/studied further to unify trainings.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be experts in the field of Cardiothoracic Surgery Critical Care Medicine to better understand the training needs of the field. Experts must have been in practice for a minimum of 5 years and have at least 50% of practice in cardiothoracic intensive care units.
* The participants will have graduated from a critical care fellowship in either an administration, education, or research role.

Exclusion Criteria:

* Participants who do not meet the exclusion criteria will be excluded due to their lack of experience in the field.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A team of experts in the field of cardiothoracic critical care anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Degree of consensus on the curriculum for training cardiothoracic critical care by first evaluating the need for the field | 12 months
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating.

SECONDARY OUTCOMES:
Degree of consensus on defining training core competencies, goals, and milestones. | 12 months
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating.
Degree of consensus on the definitions of "Scholarship", "Patient", "Safety", "Quality" | 12 months
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided